CLINICAL TRIAL: NCT00231140
Title: Randomized, Open, Parallel Group Study for the Evaluation of an Oral Dose of 100 mg Thalidomide and Subsequent Dose Escalation of 400 mg Thalidomide in Combination With Riluzole in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Pilot-Study of Thalidomide in Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THL-ALS01
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS, motor neuron disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Thalidomide; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Thalidomide (drug)

SUMMARY:
Neuroinflammation has recently emerged as a significant contributor to motor neuron damage. ALS tissue is characterized by inflammatory changes that are observed in both sporadic and familial ALS and in the ALS superoxide dismutase 1 (SOD1) transgenic mouse model. They include an accumulation of large numbers of activated microglia and astrocytes.

Proinflammatory cytokines, such as tumor necrosis factor (TNF-), are robustly upregulated in ALS. The receptor for tumor necrosis factor- (TNF-R1) is elevated at late presymptomatic as well as symptomatic phases of disease. TNF acts as a principal driver for neuroinflammation in ALS, while several co-stimulating cytokines and chemokines act to potentiate the TNF effects [4-6].

We propose an investigational therapy of ALS with oral administration of thalidomide. The rationale for this study is based on the anti-inflammatory properties of thalidomide through the modulation of inflammatory cytokines such as TNF. The primary aim of the trial is to determine whether treatment with thalidomide is safe and well tolerated in conjunction with riluzole and whether patients with ALS can tolerate daily doses of up to 400 mg. The trial is designed as feasibility study in planning for a larger phase IIb/III trial of efficacy.

DETAILED DESCRIPTION:
Study drug will be provided as 50 mg tablets. Patients will be instructed to take 2 tablets orally once a day during the evening at least 60 minutes after a meal. Thalidomide will be administered starting at 100 mg (Group 1) for 6 weeks. Thereafter, the dose will be increased every week by 50mg until reaching the dose of 400 mg/day. This treatment is continued for 12 weeks. Thalidomide is administered in conjunction with the standard treatment of riluzole (100mg/day).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 25 and 80 years
* female patients who are either postmenopausal for at least 24 month or who are willing and able to practice the methods of contraception following the Pharmion-Risk Managment Program (PRMP)
* Male patients who are willing and able to practice the methods of contraception along with their female partners of childbearing potential following the PRMP
* Clinical diagnosis of probable and definite ALS
* Sporadic or familial ALS
* Onset of pareses for no more than 4 years
* Vital capacity equal to or more than 65% of the predicted value
* Treatment with riluzole 100mg/day
* Patients who are willing to give informed consent

Exclusion Criteria:

* pregnancy or breast feeding
* female patients who are unwilling or unable to practice the methods of contraception following the Pharmion-Risk Managment Program (PRMP)
* Male patients who are willing and able to practice the methods of contraception along with their female partners of childbearing potential following the PRMP
* Patients unlikely to comply with the PRMP and other study requirements
* Patients with significant sensory abnormalities, dementia, uncompensated medical illnesses and psychiatric disorders
* Laboratory abnormalities consistent with clinically significant cardiovascular, respiratory, haematological, metabolic, hepatic and renal disease
* Infectious disease including HIV, hepatitis B and C
* monoclonal gammopathy of unknown significance (MGUS)
* History of substance abuse within the past year
* History of recurrent thrombosis
* Continuous non-invasive ventilation (ventilation-free interval equal to or less than 2 hours daily)
* Tracheotomy and invasive ventilation
* Treatment with investigational drug within 3 months prior to screening
* patients with clinically signifikant sensory polyneuropathy (inflammatory neuropathy cause and treatment sensory sum score - ISS ≥ 2)
* patients with sleep disorder (Epworth Sleeping Scale-ESS ≥ 10)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-12; Study Completion 2006-08

PRIMARY OUTCOMES:
to evaluate the long-term safety and tolerability of thalidomide
to compare the total number of adverse events (AE), abnormal laboratory tests, and number of patients who completed the study between groups

SECONDARY OUTCOMES:
to evaluate the clinical effect of two oral doses of the thalidomide on the rate of functional decline in ALS patients measured by the ALS Functional Rating Scale-revised (ALS-FRS-R) over a 24 week treatment period
to investigate the effects of thalidomide on pulmonary function (forced vital capacity) over a 24 week treatment period
to evaluate the sleep quality and somnolence using the Epworth Sleeping Scale: ESS ≥ 18
to evaluate the frequency and severity of sensory neuropathy using the inflammatory neuropathy cause and treatment sensory sum score - ISS ≥ 4
to evaluate the frequency of thrombotic events
to determine the number of patients who require continuous non-invasive ventilation or invasive ventilation
to determine the number of patients who require percutanous endoscopic gastrostomy (PEG)
to evaluate the survival time or the time point until invasive ventilation is started

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, MD, Study Chair — Charité University Hospital, Berlin, Germany
Locations (1):
- Charite University Hospital, Berlin, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Meyer T, Maier A, Borisow N, Dullinger JS, Splettstosser G, Ohlraun S, Munch C, Linke P. Thalidomide causes sinus bradycardia in ALS. J Neurol. 2008 Apr;255(4):587-91. doi: 10.1007/s00415-008-0756-3. Epub 2008 Apr 21. PMID 18425621
- See also: Related Info — http://www.als-charite.de